CLINICAL TRIAL: NCT05912192
Title: The Efficacy Of Elonide Nasal Corticosteroids In Managing Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: HOE pharmaceuticals Sdn. Bhd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF-2021-421
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elonide Nasal Spray (Experimental): Elonide is generic nasal spray Dose: 50 mcg/dose mometasone furoate 140 sprays per nasal spray One pump for both nostrils twice daily
  Interventions: Drug: Elonide Nasal Spray
- Nasonex Nasal Spray (Active Comparator): Nasonex Aqueous Nasal Spray Dose: 50 mcg/dose mometasone furoate 140 sprays per nasal spray The usual recommended dose for prophylaxis and treatment is two sprays (50 micrograms/spray) in each nostril once daily (total dose 200 micrograms) One pump for both nostrils twice daily
  Interventions: Drug: Nasonex Nasal Spray
- Normal Saline (Placebo Comparator): Placebo used is 0.9% sodium chloride Dose: 50 mcg/dose of 0.9% sodium chloride One pump for both nostrils twice daily
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Elonide Nasal Spray — 50mcg/dose One puff for each nostrils twice daily
  Other Names: Elonide
  Arms: Elonide Nasal Spray
Drug: Nasonex Nasal Spray — 50mcg/dose One puff for each nostrils twice daily
  Arms: Nasonex Nasal Spray
Drug: Normal saline — 50mcg/dose of 0.9% sodium chloride One puff for each nostrils twice daily
  Other Names: Placebo
  Arms: Normal Saline

SUMMARY:
The aim of this clinical study is to compare the efficacy of Elonide Nasal Spray to Nasonex Nasal Spray and Placebo (non-active ingredient) in the management of allergic rhinitis.

There are two hypotheses of this study:

1. Elonide nasal spray is same efficacy to Nasonex nasal spray.
2. Elonide nasal spray is more efficient to placebo.

DETAILED DESCRIPTION:
There are several objectives of the study:

1. To compare the efficacy of Elonide to Nasonex and Placebo in treating allergic rhinitis via Quality of life assessments and nasal airflow improvements.
2. To compare the efficacy of Elonide to Nasonex and Placebo in treating allergic rhinitis via symptomatics improvement.
3. To assess the side effect of Nasal spray given.

Patients who meet the criteria to join the study will be randomized in a double-blind manner (patients and investigators). Patients will be given information about the study and consent form, patients will be randomized to 3 treatment group(Elonide, Nasonex, Placebo). Patients will be evaluated before and after treatment in one month time. Patients will be advised to use the nasal spray twice daily.

ELIGIBILITY:
Inclusion Criteria:

* All adults patients 18 years and above
* Newly diagnosed mild, moderate to severe, intermittent and persistent allergic rhinitis
* Positive skin prick test or serum Immunoglobulin E

Exclusion Criteria:

* Patients who have been on allergic rhinitis treatment
* Below 18 years old
* Patients diagnosed with asthma or immunodeficiency diseases
* Pregnancy
* Other concomitant rhinology disease
* Smokers
* Severe deviated nasal septum

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Symptoms Score on Allergic Rhinitis at Week 4 | Baseline and week 4
  The Visual Analogue Score (VAS) is a validated, self-reported instrument assessing average scoring of overall allergic rhinitis symptoms in the last 7 days period from treatment date. Possible score range from 0 (no symptoms) to 100 (worst possible symptoms). Maximum number of change from baseline indicate improvement of symptoms.
  Change= (Baseline score - Week 4 score)
Mean difference from Baseline in Quality of Life Questionnaire on several domains at Week 4 | Baseline and week 4
  Rhinoconjunctivitis Quality of Life Questionnaire (RQOLQ) contains several domains score to access patient quality of life for a 7 days period from treatment date. The domains include activities, sleep, non-hay symptoms, practical problems, nasal symptoms, eye symptoms and emotional. Possible scoring from 0 (not trouble) to 6 (extremely troubled).
  Change= (Baseline score - Week 4 score)
Change from Baseline in Total Nasal Resistance while normal breathing at Week 4 | Baseline and week 4
  Total Nasal Resistance is performed using Rhinomanometry device that provides a functional measure if pressure during a breathing cycle. Normal values for total nasal resistance is below 0.2 and to 0.3 Pa cm3/s. Worst case will be higher than 0.3 Pa cm3/s indicate nasal obstruction.
  Change= (Baseline score - Week 4 score)

SECONDARY OUTCOMES:
Adverse effect of Nasal Spray | Baseline to week 4
  Any kind of side effect experience by patients in the period of using nasal spray

CONTACTS AND LOCATIONS:
Overall Officials: Hardip Singh Gendeh, Principal Investigator — Department of Otorhinolaryngology, Faculty of Medicine, Universiti Kebangsaan Malaysia
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery, Faculty of Medicine, Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in allergic rhinitis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data can be assess 6 months after publication
Access Criteria: Access to trial IPD can be access by qualified researchers engaging in independent scientific research.